CLINICAL TRIAL: NCT02618798
Title: Association of Hepatic Venous Pressure Gradient With Platelet Activation in Chronic Liver Disease
Brief Title: Hepatic Venous Pressure Gradient and Platelet Activation in Chronic Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sibylle Pramhas, M.D., Medical University of Vienna
Other Study IDs: HVPG_Platelets_Version_4.0
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Liver Disease
Keywords: chronic liver disease; CLD; platelet function

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum Plasma Platelet pellet
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Thrombosis may be crucial in driving the progression of fibrosis in chronic liver disease (CLD). The potential role of platelets and platelet activation in this process is unclear. Platelets participate in inflammation by secretion of pro-inflammatory mediators which may advance hepatic fibrosis. Hepatitis B virus transgenic mice, developed significantly smaller necroinflammatory foci and their serum ALT levels were 80% lower, if they were pre-treated with anti-platelet antibodies. Sinusoidal aggregation of activated platelets also occurs in chronic hepatitis C in humans. It may contribute to thrombocytopenia observed in CLD. Platelet activation is generally believed to be compromised in CLD. However, there is data suggesting that CLD may even be associated with an enhancement of platelet activation. Measurement of hepatic venous pressure gradient (HVPG) constitutes the most common method for estimation of portal venous pressure. HVPG is significantly correlated with histological indices of CLD progression.

Study hypotheses:

1. HVPG as a marker for advancement of hepatic fibrosis and progression of CLD is associated with an increase in platelet activation.
2. Platelet activation and function is not generally compromised in CLD. Comparison of platelet function in CLD to a control group of healthy volunteers is intended to clarify whether CLD leads to a manifest platelet dysfunction

Methods: Study design is observational. 100 patients with CLD of various origins (viral, alcoholic, cholestatic) scheduled for routine HVPG measurement will be enrolled. 30 healthy volunteers will donate blood as a control group. Platelet function and activation will be evaluated by multiple electrode aggregometry (primary outcome variable area under the curve (AUC). Plasma levels of P-selectin (ELISA), PFA (Platelet Function Analyzer) 100™ parameters (EPI-CT and ADP-CT), percentage of P-selectin, GPIIb/IIIa, thrombin receptor positive platelets after stimulation (flow-cytometry) will constitute secondary outcome parameters. Plasmatic coagulation will be evaluated by rotational thrombelastometry (ROTEM). Platelet count and routine coagulation parameters will be monitored. HVPG measurement by hepatic vein catheterization and patient blood sampling will be carried out via the internal jugular vein. Blood sampling in volunteers will be performed via the antecubital vein

Study Rationale: If higher levels of platelet activation are associated with increased HVPGs, this would provide an insight into the pathogenesis of CLD. It would also point toward a possible benefit of anti-platelet therapy in CLD. Verification of platelet dysfunction in CLD is relevant to clinical practice in anaesthesiology and intensive care as procedures are often postponed in CLD-patients for fear of bleeding complications. CLD patients may also receive prophylactic platelet concentrates prior to interventions which is costly, fraught with risk of bacterial infection and may be unnecessary in the absence of platelet dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed chronic liver disease (CLD), alcoholic, viral, cholestatic.
* CHILD-PUGH Stage A, B, C, and non-cirrhotics
* Planned routine measurement of HVPG.
* Age: 19 years or older

Exclusion Criteria:

* Impaired kidney function (Creatinine > 1.3mg/dl)
* Platelet count < 50,000/µl
* Participation in a clinical trial in the 3 weeks preceding the study
* IFN-therapy within 6 months of inclusion into the study.
* Use of anti-thrombotic or anticoagualant medication
* Pregnancy
* Intra or extra-hepatic malignancy
* Haemostatic diseases other than cirrhosis
* Current abuse of alcohol (Abstinence from alcohol for at least 6 weeks preceding the study is required)

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from chronic liver disease scheduled for routine measurement of the hepatic venous pressure gradient (HVPG).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Multiple electrode aggregometry (MEA) parameter area under the curve (AUC) | Single measurement within study duration of two years

SECONDARY OUTCOMES:
MEA parameters velocity (AU/min) | Single measurement within study duration of two years
Aggregation (AU) | Single measurement within study duration of two years
Percentage (%) of P-selectin positive platelets | Single measurement within study duration of two years
  FACS
Percentage (%) GPIIa/IIIb receptor positive platelets | Single measurement within study duration of two years
  FACS
Percentage (%) thrombin receptor positive platelets | Single measurement within study duration of two years
  FACS
P-selectin plasma level | Single measurement within study duration of two years
Serotonin plasma level | Single measurement within study duration of two years
Rotational thrombelastometry parameter: CT (coagulation time) (seconds) | Single measurement within study duration of two years
Rotational thrombelastometry parameter: CFT (clot formation time) (seconds) | Single measurement within study duration of two years
Rotational thrombelastometry parameter: MCF (maximum clot firmness) (mm) | Single measurement within study duration of two years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Special Anesthesia and Pain Therapy, Medical University of Vienna, AKH Vienna, Vienna, Vienna, Austria